CLINICAL TRIAL: NCT03173404
Title: Benefits of Hysteroscopy Prior to Performing a Cycle of in Vitro Fertilization/Intracytoplasmic Sperm Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3913
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Sterility
MeSH Terms: conditions — Infertility | interventions — Hysteroscopy

STUDY DESIGN:
Intervention Model Description: Randomized open-label clinical trial. Women scheduled for their first or second IVF/ICSI cycle and with no abnormality detected in transvaginal ultrasound examination, were randomized to two groups.
  In the first group (group I): 31 patients underwent hysteroscopy examination before IVF cycle.
  The second group (group II): 37 patients underwent direct cycle without previous hysteroscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients underwent hysteroscopy examination before IVF cycle.
  Interventions: Procedure: Hysteroscopy
- Group II (No Intervention): Patients underwent direct IVF cycle without previous hysteroscopy.

INTERVENTIONS:
Procedure: Hysteroscopy — The hysteroscopy is the visualization of the cervical canal and uterine cavity with a camera. Patients randomized to group I underwent hysteroscopy prior to the IVF cycle.
  Arms: Group I

SUMMARY:
This is a prospective randomized open-label trial. Women scheduled for their first or second in-vitro fertilization/intracytoplasmatic Sperm Injection (IVF/ICSI) cycle and with no abnormality detected in transvaginal ultrasound examination, were randomized to two groups. In the first group (group I) 31 patients underwent hysteroscopy examination before IVF cycle while in the second group (group II) 37 patients underwent direct cycle without previous hysteroscopy

DETAILED DESCRIPTION:
This is a prospective randomized open-label trial. Women scheduled for their first or second IVF/ICSI cycle and with no abnormality detected in transvaginal ultrasound examination, were randomized to two groups. In the first group (group I) 31 patients underwent hysteroscopy examination before IVF cycle while in the second group (group II) 37 patients underwent direct cycle without previous hysteroscopy. Then IVF cycle was performed with habitual protocol. Beta Corionic Gonatropic hormone (BhCG) test two weeks after embryo transfer was done. If test was positive, patients were followed up for detection pregnancy by transvaginal ultrasound two weeks later. Another transvaginal ultrasound at 12 weeks of gestation was done to confirm ongoing pregnancy. Biochemical pregnancy, implantation, on-going pregnancy and livebirth rates were compared in both groups.

Miscarriage, complications rate and hysteroscopy tolerability were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women with infertility / primary infertility.
* Women who are about to start an IVF/ICSI cycle with their own eggs.
* Age greater than or equal to 18 years and less than or equal to 40 years.
* Women in whom a multiple follicular development will be developed with a short protocol with antagonists or long with agonists, and starting dose of gonadotropins according to clinical criteria.
* Women with uterine ultrasound without endometrial pathology

Exclusion Criteria:

* Ovarian reserve: Antimullerian hormone <0.5 ng / dl or Count of antral follicles <5 between both ovaries.
* Myomatous uterus: presence of> 2 myomas> 4cm or that deform uterine cavity.
* Uterine malformations.
* Body mass index (BMI) <18 or> 30.
* Polycystic ovarian syndrome: according to European Society of Human Reproduction and Embryology (ESRHE)/Rotterdam 2003 criteria.
* Moderate-severe endometriosis.
* Background or presence of pelvic inflammatory disease.
* Hydrosalpinx not excised or occluded.
* Hyperprolactinemia, defined as prolactin levels greater than 50 ng / ml.
* Diagnostic history of endometrial hyperplasia.
* Severe male factor: severe oligoasthenoteratozoospermia with a sperm cell count (REM) <100,000 spermatozoa / ml.
* Impossibility to apply the treatments provided by the study in the terms established by the protocol.
* Contraindication for the use of any of the treatments provided in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients included in the study must be female with uterus.
Enrollment: 75 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percentage of biochemical, clinical, on-going pregnancy and livebirth of IVF treatment | 12 months
  Percentage of biochemical, clinical, on-going pregnancy and livebirth of IVF treatment comparing both groups.

SECONDARY OUTCOMES:
Percentage of endocervical canal and uterine cavity pathology and the impact of treatment of these pathologies. | 12 months
  Percentage of endocervical canal and uterine cavity pathology and the impact of treatment of these pathologies in the rate of pregnancy and livebirth.
Rate of hysteroscopy tolerance | 1 month.
  The tolerance of the procedure was evaluate in the patients randomized to the group I of the study.
Hysteroscopy complication rate. | 2 months
  We evaluate the complication of the hysteroscopy during and after the procedure. Includes blooding, infections, uterine perforation, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No